CLINICAL TRIAL: NCT05163379
Title: EARLY MOBILIZATION OF INTUBETED PATIENTS IN THE INTENSİVE CARE UNİT AND THE EFFECTS OF EARLY MOBILIZATION ON RESPIRATORY PATTERN AND PATIENT HEMODYNAMICS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gürkan ÇAMOK, Nursing Graduate Student, Okan University
Other Study IDs: GURKANCAMOK
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Intensive Care Unit Acquired Weakness; Intensive Care, Intubated Patient, Early Mobilization, Mobilization, Respiratory Pattern

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INTENSIVE CARE PATIENTS: EARLY MOBILIZATION OF INTUBE PATIENTS
  Interventions: Other: MOBILIZATION

INTERVENTIONS:
Other: MOBILIZATION — EARLY MOBILIZATION OF INTUBE PATIENTS AND ITS EFFECTS OF MOBILIZATION

SUMMARY:
The present study was carried out as a quasi-experimental study in order to examine the effects of early mobilization of intubated patients in the intensive care unit and the effects of early mobilization on respiratory pattern and patient hemodynamics. The sample of the study consisted of 25 intubated patients monitored in the intensive care unit at in a private hospital between May 2020 and July 2021. Ethics committee approval and study permission were obtained from the hospital before starting the data collection process. Research data, descriptive data collection form, Richmond- Agitation Sedation Scale (RASS) scale, Muscle Strength Testing (Oxford Scale) and with the mobilization of the patients 45 minute in 30-60 minute including the preparation process, (1st Stage Semi Fowler position, 2nd Stage bedside sitting position, 3rd Stage in the bedside sitting position after mobilization) were registered in the Early Mobilization Follow-up Form and collected. Number and percentage calculations, repeated measurement ANOVA and Post Hoc Sheffe, LSD test analyzes were utilized in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Hemodiamic stability (OCD >60, OCD <120, respiratory rate <35, SpO2 >90),
* Areas of >3/5 (Oxford scale) and above on the lower limbs with areas of secure support,
* The patient scores 0 (awake and calm) on the Richmond Agitation Sedation Scale (RASS),
* PaO2 / FiO2 ≥300,
* Body temperature below 38 degrees,
* Platelet count ≥20,000 cells / mm3,
* Having blood sugar of 60-360 mg/dl,
* Having arterial monitoring,
* Patient with 30% FiO2 due to mechanical ventilator,
* Those with mechanical ventilator-dependent ventilation method (mode) PASB,
* Patient with a PEEP value of 5 due to mechanical ventilator,
* Patient with a PASB value of 10 connected to a mechanical ventilator,
* A sample accepted by the patient who voluntarily agreed to participate in the study was approximated from the patient.

Exclusion Criteria:

* Patients under the age of 18,
* Those with hemodynamic instability (OCD <60 mmHg, OCD >120 mmHg, breath rate >35, SpO2 <90),
* Those who do not have secure unsupported sitting balance and have a score of >3/5 (Oxford scale) in the lower limbs,
* Patients whose Richmond agitation sedation scale (RASS) is between +1 and +4 points, and patients with a score between -1 and -5,
* Those with arrhythmia,
* Patients without arterial monitoring,
* Patients whose FiO2 percentage is not 30% in patients on mechanical ventilator,
* Patients who do not have ventilation method (mod) PASB in patients on mechanical ventilator,
* Patients who do not have a PEEP value of 5 in patients on mechanical ventilators,
* Patients who do not have a PASB value of 10 in patients on mechanical ventilators,
* Those with neurological and orthopedic contraindications,
* Patients who could not get approval from the relatives of the patients who did not accept to participate in the study were excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: INTUBE PATIENTS IN ICU
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
EARLY MOBILIZATION OF INTUBE PATIENTS AND THE EFFECTS OF EARLY MOBLIZATION ON RESPIRATORY PATTERN AND PATIENT HEMODYNAMICS | ONE DAY
  HEMODYNAMIC EFFECTSRESPIRATORY PATTERN, BLOOD GAS ANALYSISZ

CONTACTS AND LOCATIONS:
Locations (1):
- Gürkan ÇAMOK, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
all of

REFERENCES:
- [Background] Green M, Marzano V, Leditschke IA, Mitchell I, Bissett B. Mobilization of intensive care patients: a multidisciplinary practical guide for clinicians. J Multidiscip Healthc. 2016 May 25;9:247-56. doi: 10.2147/JMDH.S99811. eCollection 2016. PMID 27307746
- Available data/document: Study Protocol — https://khgmekodemedb.saglik.gov.tr/Eklenti/23273/0/fizik-tedavi-ve-rehabilitasyon-islemleri-degerlendirme-olcekleripdf.pdf